CLINICAL TRIAL: NCT00543712
Title: A Phase II, Open-Label, Multicenter Study of the Efficacy and Safety of Single-Agent PRO95780 in Patients With Advanced Chondrosarcoma
Brief Title: A Study of PRO95780 in Patients With Advanced Chondrosarcoma (APM4171g)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy not evident in this population.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: APM4171g
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Chondrosarcoma
Keywords: Sarcoma; synovial sarcoma; APM4171g
MeSH Terms: conditions — Chondrosarcoma; Sarcoma; Sarcoma, Synovial | interventions — drozitumab

ARMS (1):
- PRO95780 (Experimental)
  Interventions: Drug: PRO95780

INTERVENTIONS:
Drug: PRO95780 — Intravenous repeating dose

SUMMARY:
This is a multicenter, open-label, Phase II trial designed to evaluate the efficacy and safety of PRO95780 when given as a single agent in patients with advanced chondrosarcoma. Up to 90 patients with confirmed chondrosarcoma will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document
* Age ≥ 18 years
* Histologic diagnosis of chondrosarcoma, verifiable after enrollment
* Measurable disease
* Previously treated or incurable disease without options for standard of care therapy
* ECOG performance status of 0-2
* Life expectancy of > 3 months
* For patients of reproductive potential (males and females), use of reliable means for contraception (e.g., contraceptive pill, intrauterine device [IUD], physical barrier) throughout the trial and for 1 year following their final exposure to study treatment

Exclusion Criteria:

* Systemic therapy or radiotherapy within 4 weeks prior to Day 1
* Prior therapy with agents targeting the DR5 apoptosis pathway
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Other invasive malignancies within 5 years prior to Day 1
* Known active brain metastases
* Uncontrolled intercurrent illness, including but not limited to ongoing or active infection requiring parenteral antibiotics at enrollment
* Clinically significant, symptomatic cardiovascular disease, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia, Grade II or greater peripheral vascular disease, or history of major heart surgery within 6 months of Day 1, or any situation that would likely limit compliance with study requirements
* Known to be positive for hepatitis C or hepatitis B surface antigen
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk for treatment complications
* Use of anticoagulation therapy
* Participation in clinical trials or undergoing other investigational procedures within 30 days prior to Day 1
* Pregnancy or breast feeding
* Known sensitivity to any of the products administered during the study
* Any disorder that compromises the ability of the patient to give written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05-31 (Actual); Primary Completion 2008-05-05 (Actual); Study Completion 2008-05-05 (Actual)

PRIMARY OUTCOMES:
Adverse events
Change in vital signs before and after PRO95780 infusions; clinical laboratory evaluations
Objective response

SECONDARY OUTCOMES:
Duration of objective response
Progression-free survival
Overall survival
Pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Skettino, M.D., Study Director — Genentech, Inc.
Locations (4):
- United States (3):
  - Sarcoma Oncology Center, Santa Monica, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Centre, Melbourne, Australia